CLINICAL TRIAL: NCT03449940
Title: Penile Fracture: A Prospective Randomized Study Comparing Erectile Function at 12 Months After Immediate Degloving Repair Versus Delayed Localized Repair
Brief Title: Penile Fracture: A Comparison of Erectile Function After Immediate Repair Versus Delayed Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Jamaica (Other)
Collaborators: University Hospital of the West Indies (Other)
Responsible Party: Principal Investigator, Dean Wong, Principal Investigator, Ministry of Health, Jamaica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4200
Record Dates: First submitted 2018-02-11; First posted 2018-02-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Erectile Dysfunction
Keywords: Penile fracture; Delayed; Localized; Repair
MeSH Terms: conditions — Erectile Dysfunction | interventions — Lidocaine; Anesthesia, Local; Ceftriaxone; Anti-Bacterial Agents; Diclofenac; Analgesics

STUDY DESIGN:
Intervention Model Description: A block randomization sequence was created and cases were allocated 1:1 to either immediate repair (group 1) or delayed repair (group 2). Allocation sequence numbers were kept concealed in sequentially numbered folders and access was only granted to the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate repair (group 1) (Active Comparator): Penile explorations were done within 24 hours of presentation, under general or spinal anaesthesia.
  1g Ceftriaxone IV was given.
  Incision-- Subcoronal, circumferential & degloving.
  Repair-- Continuous technique with inverted knots using 3-0 polyglactin suture.
  All patients were discharged from hospital within 24 hours.
  Interventions: Procedure: Immediate repair; Drug: Ceftriaxone
- Delayed repair (group 2) (Active Comparator): Patients were not admitted; instead they were discharged from hospital and given an elective surgery date. Oral Diclofenac Sodium 50mg was prescribed to be taken as needed and instructions to abstain from any sexual activity.
  In an ambulatory setting, surgery was done 7 - 10 days later.
  1g Ceftriaxone IV was given.
  Local anaesthesia (dorsal penile nerve block): 1% Lidocaine 10cc was given.
  Incision--- 2 - 3cm localized incision over the site of the "rolling" sign.
  Repair--- Continuous technique with inverted knots using 3-0 polyglactin suture.
  Interventions: Procedure: Delayed repair; Drug: Lidocaine; Drug: Ceftriaxone; Drug: Diclofenac Sodium

INTERVENTIONS:
Procedure: Immediate repair
  Arms: Immediate repair (group 1)
Procedure: Delayed repair
  Arms: Delayed repair (group 2)
Drug: Lidocaine — 10cc of Lidocaine 1% is used to inject at the base of the penis for a dorsal penile nerve block for the localized repair.
  Other Names: Local Anaesthesia
  Arms: Delayed repair (group 2)
Drug: Ceftriaxone — Pre-operative antibiotic given to all patients. Ceftriaxone 1g is administered intravenously.
  Other Names: Antibiotic
Drug: Diclofenac Sodium — Oral Diclofenac Sodium 50mg tablet is prescribed to be taken as needed up to a maximum of three times daily until the penis is repaired.
  Other Names: Analgesic
  Arms: Delayed repair (group 2)

SUMMARY:
To prospectively compare erectile function at 12 months, utilizing the abbreviated International Index of Erectile Function-5 (IIEF-5) score, for men treated with an immediate repair versus a delayed repair.

DETAILED DESCRIPTION:
This was a prospective randomized study conducted at 2 tertiary level institutions in Jamaica, the University Hospital of the West Indies (UHWI) and the Kingston Public Hospital (KPH). All cases of penile fracture were recruited from the emergency room (ER) of both hospitals between the period January 2015 to January 2017 and all patients were over 18 years of age.

Information on demographics, length of time since the injury, mechanism of injury and risk factors for erectile dysfunction (Diabetes mellitus, Hypertension, Dyslipidemia, Smoking) was collected. Erectile function was objectively assessed utilizing the abbreviated International Index for Erectile Function-5 (IIEF-5), and scores at initial presentation were taken to represent the premorbid erectile function.

A block randomization sequence was created and cases were allocated 1:1 to either immediate repair (group 1) or delayed repair (group 2). Allocation sequence numbers were kept concealed in sequentially numbered folders and access was only granted to the principal investigator.

For Group 1 (Immediate repair)

Patients were admitted to hospital and underwent emergency repair via a subcoronal circumferential degloving approach.

For Group 2 (Delayed repair)

Patients were not admitted. Instead, they were discharged from hospital and given an elective surgery date 7 - 10 days after the injury. Oral Diclofenac Sodium 50mg was prescribed to be taken as needed and instructions to abstain from any sexual activity.

All patients were then re-examined at 6 weeks for quality assurance. They were then instructed that resumption of sexual activity would be safe.

Routine clinic visits were scheduled at 3 months, 6 months, and 12 months. IIEF-5 scores were obtained from all patients at 12months.

ELIGIBILITY:
Inclusion Criteria:

* Men with penile fracture presenting to the emergency room

Exclusion Criteria:

* Suspicion of concomitant urethral injury (blood at the meatus, gross/microscopic haematuria, urinary retention)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Erectile function | 12 months
  The International Index of Erectile Function (IIEF-5) is recorded as a total score. It is measured by a self-reported questionnaire with 5 domains, with each domain consisting of 5 options. The score ranges from 5 to 25, with 5 being the lowest score (severe erectile dysfunction) and 25 being the best score (maximal erection).

SECONDARY OUTCOMES:
Penile nodule | 12 months
  The penis is examined and palpated for the presence of nodule formation at the fracture repair site. It is recorded as "present" or "not present".
Penile pain during sexual intercourse | 12 months
  The patient is asked if there is pain in the penis during sexual intercourse. It is recorded as "present" or "not present".
Penile curvature | 12 months
  The patient is asked if there is an acquired curvature of the erect penis. It is recorded as "present" or "not present".
Patient satisfaction | 12 months
  The Surgical Satisfaction Questionnaire (SSQ-8) is administered. There are 8 questions with 5 possible options in each domain. The questionnaire results are recorded as descriptive terms for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Morrison, DM(Urol) PhD, Study Director — University of the West Indies
Locations (2):
- Jamaica (2):
  - Kingston Public Hospital, Kingston
  - University Hospital of the West Indies, Kingston

IPD SHARING:
Plan to Share IPD: No